CLINICAL TRIAL: NCT04061590
Title: A Phase 2 Study of Neoadjuvant Pembrolizumab-Based Combination Immunotherapy in the Treatment of Early Stage Non-Small Cell Lung Cancer
Brief Title: Pembrolizumab With or Without Chemotherapy Before Surgery in Treating Patients With Stage I-IIIA Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Matthew Gubens, MD, Principal Investigator, University of California, San Francisco
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19702; NCI-2019-04763 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; pembrolizumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (pembrolizumab) (Experimental): Patients receive 200mg pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery within 4 weeks following study treatment.
  Interventions: Biological: Pembrolizumab; Procedure: Therapeutic Conventional Surgery
- Cohort B (pembrolizumab, cisplatin pemetrexed) (Experimental): Patients receive 200mg pembrolizumab IV over 30 minutes and chemotherapy (cisplatin/pemetrexed) IV on day 1. Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery within 4 weeks following study treatment.
  Interventions: Drug: Cisplatin; Biological: Pembrolizumab; Drug: Pemetrexed; Drug: Pemetrexed Disodium; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Cohort B (pembrolizumab, cisplatin pemetrexed)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate
  Arms: Cohort B (pembrolizumab, cisplatin pemetrexed)
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt
  Arms: Cohort B (pembrolizumab, cisplatin pemetrexed)
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase II trial studies how well pembrolizumab with or without chemotherapy works when given before surgery in treating patients with stage I-IIIA non-small cell lung cancer. Immunotherapy with pembrolizumab, may induce changes in body?s immune system and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as cisplatin and pemetrexed, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pembrolizumab with or without chemotherapy may shrink the cancer prior to surgery and decrease the likelihood of the cancer returning following surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the impact of neoadjuvant pembrolizumab-based combination therapy on the composition, phenotype, and function of tumor-infiltrating immune cells (TIICs) in patients with early stage non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of neoadjuvant pembrolizumab alone and in combination with chemotherapy as measured by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0.

II. To determine the clinical efficacy of neoadjuvant pembrolizumab alone and in combination with chemotherapy.

EXPLORATORY OBJECTIVES:

I. To explore the relationship between changes in TIICs and clinical efficacy in patients with early stage NSCLC treated with neoadjuvant pembrolizumab-based combination therapy.

II. To characterize changes in the frequency and number of circulating immune cells induced by neoadjuvant pembrolizumab-based combination therapy in patients with early stage NSCLC.

III. To determine the impact of neoadjuvant pembrolizumab-based combination therapy on the composition and phenotype of the tumor microenvironment (including tumor and stromal cells) in patients with NSCLC.

III. To determine the change in T cell repertoire within the tumor and blood induced by neoadjuvant pembrolizumab-based combination therapy in patients with early stage NSCLC.

IV. To explore molecular profiles to identify potentially predictive biomarkers for patients with early stage NSCLC treated with immunotherapy.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery within 4 weeks following study treatment.

COHORT B: Patients receive pembrolizumab IV over 30 minutes and chemotherapy (cisplatin/pemetrexed) IV on day 1. Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery within 4 weeks following study treatment.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC, performed on a biopsy that occurred within the last 60 days
* Computed tomography (CT) within the last 30 days showing radiographic stage I to IIIa lung cancer (mediastinal staging biopsy is allowed but not required) by the American Joint Committee on Cancer (AJCC) 8th edition
* Documentation that the patient is a candidate for surgical resection of their lung cancer by an American Board of Thoracic Surgery-certified surgeon
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by the investigator
* Adequate tissue specimens for correlative biomarker analysis. The patient should be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 8 weeks (56 days) prior to initiation of treatment on day 1. Patients for whom newly-obtained samples cannot be provided (e.g. inaccessible or patient safety concern) may submit an archived specimen only upon agreement from the principal investigator
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Resolution of all acute toxic effects of prior chemotherapy, radiotherapy or surgical procedures to NCI CTCAE version (v)5.0 grade 1
* Be willing and able to provide written informed consent for the trial
* Absolute neutrophil count (ANC) >= 1500 cells/ microlitre(uL) (within 10 days prior to the start of trial treatment)
* Platelets >= 100 000 cells/uL (within 10 days prior to the start of trial treatment)
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L (criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks) (within 10 days prior to the start of trial treatment)
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance, glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl) >= 30 mL/min for patients with creatinine levels > 1.5 x institutional ULN (within 10 days prior to the start of trial treatment)
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for patients with total bilirubin levels > 1.5 x ULN (within 10 days prior to the start of trial treatment)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 2.5 x ULN (=< 5 x ULN for patients with liver metastases) (within 10 days prior to the start of trial treatment)
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 10 days prior to the start of trial treatment)
* Activated partial thromboplastin time (aPTT)/PTT =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 10 days prior to the start of trial treatment)
* Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of trial medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Male and female patients of childbearing potential must be willing to use an adequate method of contraception as outlined, for the course of the trial through 120 days after the last dose of trial drug

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient
* Be willing to provide newly obtained tissue (core biopsy of tumor) for PD-L1 biomarker analysis and, based on the adequacy of the tissue sample quality for assessment of PD-L1 status, received permission for enrollment from the core laboratory. Repeat samples may be required if adequate tissue is not provided. Newly obtained biopsy specimens are preferable to archived samples, and formalin-fixed paraffin-embedded (FFPE) block specimens are preferred to slides. A post-treatment biopsy after pembrolizumab treatment is desirable if patient agrees

  * Collection of an archived tissue sample will also be requested available) to support evaluation of the clinical utility of PD-L1 assessment in newly obtained versus (vs.) archived tissue samples; however, a patient will not be precluded from participating in the study if an archived tissue sample is not available for collection or is otherwise insufficient for analysis

Exclusion Criteria:

* Is ineligible for an operation based on medical or oncologic contraindications to surgery
* Is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of trial treatment

  * Note: Patients who have entered the follow-up phase of an investigational trial may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
* Has any component of small cell tumor in the specimen, e.g. mixed NSCLC/small cell
* Has received prior therapy with an anti-Programmed cell death protein 1 (PD-1), anti-Programmed death-ligand 1 (PD-L1) , or anti-Programmed death-ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX-40, CD137)
* Has severe hypersensitivity >= grade 3) to pembrolizumab and/or any of its excipients
* Has a history of (non-infectious) pneumonitis / interstitial lung disease that required treatment with steroids or has current pneumonitis / interstitial lung disease that requires steroids
* Has a known history of human immunodeficiency virus (HIV) infection

  * Note: No HIV testing is required unless mandated by local health authority
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (HCV) (defined as HCV ribonucleic acid [RNA] [qualitative] is detected) infection

  * Note: No testing for hepatitis B and hepatitis C is required unless mandated by local health authority
* Has a known history of active tuberculosis (TB; Mycobacterium tuberculosis)
* Has received prior radiotherapy within 2 weeks of start of trial treatment. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Has received a live vaccine within 30 days prior to the first dose of trial drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
* Has evidence of clinically significant interstitial lung disease
* Has an active second malignancy, i.e. patient known to have potentially fatal cancer present for which he/she may be (but not necessarily) currently receiving treatment. Patients with a history of malignancy that has been completely treated, with no evidence of that cancer currently, are permitted to enroll in the trial if curative therapy has been completed, such as basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient?s participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator, including dialysis
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment
* Has had an allogeneic tissue/solid organ transplant

ADDITIONAL EXCLUSION CRITERIA For Arm B

* Has squamous cell carcinoma. Adenosquamous and adenocarcinoma with squamous features disease allowed
* Creatinine clearance < 45 ml/min as calculated by institutional standard
* Is taking any herbal/complementary oral or IV medicine within 4 weeks of first dose of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a >= 2-fold increase in the number of tumor-infiltrating immune cells (TIICs) in post- versus (vs.) pre-pembrolizumab treatment tumor specimens | Up to 2 years
  Will be summarized by descriptive statistics (median and range).

SECONDARY OUTCOMES:
Proportion of participants reporting treatment-related adverse events (AEs) | Up to 2 years
  AEs determined to be treatment-related will be assessed by using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Overall Response Rate | Up to 2 years
  Response rate is the proportion of participants with a complete response or partial response as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Clinical Benefit Rate | Up to 2 years
  Clinical benefit rate is defined as the proportion of participants with a complete response, partial response, or stable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Median Progression-Free Survival (PFS) | 12 months
  Median PFS following surgical resection is defined as the time from objective response (complete response or partial response) to the time in which a diagnosis of disease progression has occurred. Kaplan-Meier estimates will be generated and participants will be censored at 12 months.
Median Progression-Free Survival (PFS) | 24 months
  Median PFS following surgical resection is defined as the time from objective response (complete response or partial response) to the time in which a diagnosis of disease progression has occurred. Kaplan-Meier estimates will be generated and participants will be censored at 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Gubens, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No